CLINICAL TRIAL: NCT05601921
Title: Effects of High Frequency Repetitive Transcranial Magnetic Stimulation on Pain and Disability in Patients With Post-stroke Shoulder Pain
Brief Title: Repetitive Transcranial Magnetic Stimulation in Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Yagmur Aydin, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-TDU-TIPF-0013
Record Dates: First submitted 2022-10-20; First posted 2022-11-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Post-stroke Shoulder Pain
Keywords: Stroke; Shoulder pain; Repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Stroke; Shoulder Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation group (Experimental): Patients in the real stimulation group will receive rTMS treatment to the motor cortex (M1) of the affected hemisphere at a frequency of 5 Hz, once a day for 3 weeks and a total of 15 sessions. The application will be performed with Neurosoft-Neuro MS / D device. Before each session, the patient's resting motor threshold (RMT) value will be determined. RMT will be detected by obtaining a motor evoked potential of >50 μV amplitude on electromyography recording of the contralateral first dorsal interosseous muscle in at least five out of 10 stimulations to the primary motor cortex.The stimulus intensity to be used in the treatment will be set as 90% of the motor threshold for the affected motor cortex and 100% of the motor threshold for the unaffected motor cortex.One session of stimulation will last for a total of 20 minutes and a total of 1000 pulses in the form of 5 Hz stimulation.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- Sham stimulation group (Sham Comparator): Fifteen sessions of sham repetitive transcranial magnetic stimulation (rTMS) treatment will be applied to the lesional primary motor cortex. The application will be performed with Neurosoft-Neuro MS / D device. The probe of the device will be held perpendicular to the motor cortex and operated from the lowest operating power of 1, so that the device makes the same sounds as the active application.
  Interventions: Device: Sham Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive intervention that uses magnetic fields to stimulate nerve cells to improve the symptoms of a variety of disorders. In recent years, TMS studies have been conducted in many painful conditions, which are thought to have complex pain mechanisms in the pathogenesis, and its effectiveness has been reported.
  Arms: Active stimulation group
Device: Sham Repetitive transcranial magnetic stimulation — Sham Repetitive transcranial magnetic stimulation
  Arms: Sham stimulation group

SUMMARY:
Shoulder pain after stroke is one of the most common complications of stroke. Underlying mechanisms of shoulder pain after stroke still completely is not clarified. Central sensitization and neuropathic pain mechanisms are thought to play a role in the etiology of pain. Research on repetitive transcranial magnetic stimulation therapy in the treatment of pain in which somatosensory sensitization mechanisms play a role is increasing day by day. There are studies showing that application of high-frequency rTMS to the primary motor cortex provides effective pain relieving in most of painful conditions. However, data in the literature regarding the application of high-frequency rTMS in shoulder pain after stroke are very limited. There is only one clinical study related to this. More studies are needed in this area.In our study, it was aimed to examine the effects of this treatment protocol applied on the effects of pain on daily activities, upper extremity disability, anxiety, depression, range of motion and neurophysiological parameters.

DETAILED DESCRIPTION:
Stroke is one of the most common causes of disability and death in the adult population. Many complications such as depression, shoulder pain, falls, urinary system infections can develop after stroke. These complications prevent stroke rehabilitation and delay functional recovery. Hemiplegic shoulder pain is also one of the most common complications after stroke. Many possible causes underlying its development have been described; It may develop due to many pathologies such as rotator cuff lesions, biceps tendinopathy, soft tissue disorders such as myofascial pain, glenohumeral subluxation, spasticity, changes in peripheral and central nervous system activity. Many options such as joint range of motion (ROM) exercises, electrical stimulation, analgesics, intra-articular injections of corticosteroids, botulinum toxin-A injections are used in the management of pain. However, current treatment options provide limited pain relief, which causes chronic pain in many patients. This suggests that post-stroke shoulder pain is not only due to simple nociceptive stimuli from the shoulder joint, but also includes nociceptive and neuropathic mechanisms related to both the peripheral and central nervous systems. In recent years, TMS studies have been conducted in many painful conditions, which are thought to have complex pain mechanisms in the pathogenesis, and its effectiveness has been reported.In our study, it was aimed to examine the effects of this treatment protocol applied on the effects of pain on daily activities, upper extremity disability, anxiety, depression, range of motion and neurophysiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-70
* Presence of ischemic or hemorrhagic stroke confirmed by MRI
* Having a stroke for the first time
* Presence of stroke in the subacute or chronic period
* Presence of subacute or chronic shoulder pain starting after stroke and Numeric Rating Scale >4
* If the patient is receiving analgesic treatment, the pain persists despite at least one week of analgesic treatment.
* Patients who agreed to participate by signing the informed permission form.

Exclusion Criteria:

* Presence of history of surgical intervention on the shoulder joint
* Presence of history of peri/intraarticular injection into the shoulder joint
* Rotator cuff injury or tendonitis, frozen shoulder, etc. that they had diagnosed/treated before stroke
* Presence of full-thickness rotator cuff tear visualized by US
* Presence of >3 spasticity in the upper extremity defined according to the Modified Ashworth Scale
* Presence of severe cognitive impairment
* Presence of aphasia
* History of malignancy or systemic rheumatic disease
* Alcohol or drug addiction
* History of psychiatric illness such as major depression/personality disorders
* History of epilepsy or taking medication due to epilepsy
* Diagnosed with dementia
* Pregnancy and breastfeeding
* Having received TMS treatment before
* Having a clinical condition (metallic implant, cardiac pace, head trauma, cranial operation history…) that would be a contraindication for TMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Numeric Rating Scale | (1) at the beginning of the treatment, (2) at the 1st week, (3) at the 2nd week, (4) at the end of the treatment (3rd week), (5)one month after the end of the treatment
  The NRS is an 11-point numerical scale that evaluates the intensity of pain in adults from 0 to 10. 0 represents no pain and 10 represents the worst possible pain.

SECONDARY OUTCOMES:
Change from baseline in the Brief Pain Inventory - Pain on Daily Activities | (1) at the beginning of the treatment, (2) at the end of the treatment (3rd week), (3) one month after the end of the treatment
  The BPI is a two-part multidimensional pain assessment questionnaire that evaluates pain intensity and the effect of pain on daily activities (general activity, mood, walking ability, work, relationships with other people, sleep, enjoyment of life).
Change from baseline in the Quick DASH | (1) at the beginning of the treatment, (2) at the end of the treatment (3rd week), (3) one month after the end of the treatment
  It is an outcome measure developed for the evaluation of patients with upper extremity musculoskeletal disorders.
Change from baseline in the Hospital Anxiety and Depression Scale | (1) at the beginning of the treatment , (2) at the end of the treatment (3rd week)
  The hospital anxiety and depression scale (HADS) was developed to screen for depression and anxiety in hospitalized patients
Change from baseline in the shoulder joint range of motion | (1) at the beginning of the treatment, (2) at the end of the treatment (3rd week)
  Maximum painless passive range of motion values were measured as abduction adduction internal and external rotation with a goniometer in the supine position.

CONTACTS AND LOCATIONS:
Overall Officials: Ayhan Aşkın, Professor, Study Director — Izmir Katip Çelebi University; Yağmur Aydın, M.D., Principal Investigator — Izmir Katip Çelebi University
Locations (1):
- İzmir Katip Çelebi Üniversitesi, Izmir, Karabağlar / İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergen DC, Silberberg D. Nervous system disorders: a global epidemic. Arch Neurol. 2002 Jul;59(7):1194-6. doi: 10.1001/archneur.59.7.1194. PMID 12117370
- [Background] Langhorne P, Stott DJ, Robertson L, MacDonald J, Jones L, McAlpine C, Dick F, Taylor GS, Murray G. Medical complications after stroke: a multicenter study. Stroke. 2000 Jun;31(6):1223-9. doi: 10.1161/01.str.31.6.1223. PMID 10835436
- [Background] McLean DE. Medical complications experienced by a cohort of stroke survivors during inpatient, tertiary-level stroke rehabilitation. Arch Phys Med Rehabil. 2004 Mar;85(3):466-9. doi: 10.1016/s0003-9993(03)00484-2. PMID 15031834
- [Background] Kalichman L, Ratmansky M. Underlying pathology and associated factors of hemiplegic shoulder pain. Am J Phys Med Rehabil. 2011 Sep;90(9):768-80. doi: 10.1097/PHM.0b013e318214e976. PMID 21430513
- [Background] Viana R, Pereira S, Mehta S, Miller T, Teasell R. Evidence for therapeutic interventions for hemiplegic shoulder pain during the chronic stage of stroke: a review. Top Stroke Rehabil. 2012 Nov-Dec;19(6):514-22. doi: 10.1310/tsr1906-514. PMID 23192716
- [Background] Roosink M, Renzenbrink GJ, Geurts AC, Ijzerman MJ. Towards a mechanism-based view on post-stroke shoulder pain: theoretical considerations and clinical implications. NeuroRehabilitation. 2012;30(2):153-65. doi: 10.3233/NRE-2012-0739. PMID 22430581
- [Background] Choi GS, Chang MC. Effects of high-frequency repetitive transcranial magnetic stimulation on reducing hemiplegic shoulder pain in patients with chronic stoke: a randomized controlled trial. Int J Neurosci. 2018 Feb;128(2):110-116. doi: 10.1080/00207454.2017.1367682. Epub 2017 Oct 2. PMID 28805107